CLINICAL TRIAL: NCT05922995
Title: A Single Center, Open Label Prospective Observational Pilot Study to Evaluate the Effects of Tasimelteon in Participants With REM Behavior Disorder (RBD)
Brief Title: The Effects of Tasimelteon in Participants With REM Behavior Disorder (RBD)
Acronym: RBD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study will not longer be done. Terminated due to sponsor noncompliance.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Vanda Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Pavlova, Milena,M.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001873
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: REM Behavior Disorder
Keywords: REM behavior disorder; RBD; REM disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Phase (Experimental): Tasimelteon will be administered in 20 mg capsules on a nightly basis for 4 weeks during the treatment phase.
  Interventions: Drug: Tasimelteon

INTERVENTIONS:
Drug: Tasimelteon — 20 mg capsules taken on a nightly basis
  Other Names: Hetlioz

SUMMARY:
To assess the effects of a daily single oral dose of 20 mg tasimelteon compared to baseline on events of dream enactment on patients with REM Behavior Disorder, as measured by a daily log.

To assess the effects of 20 mg tasimelteon compared to baseline on insomnia= symptoms, as measured by validated questionnaires (Insomnia Severity Index [ISI], Pittsburgh Sleep Quality Inventory [PSQI], Epworth Sleepiness Scale [ESS], Clinical Global Impression of Change Scale (CGI-C), Patient Global Impression of Change Scale (PGI-C)) as well as rest/activity pattern from actigraphy.

* To assess the effects of 20 mg tasimelteon on patients who have a reduced or aberrant melatonin secretion compared to normal secretion by measuring salivary DLMO at baseline and correlating with the degree of change in RBD symptoms by end of the study.
* To assess for any role a patient's unique genome may play in their response to tasimelteon; obtained via whole genome sequencing.
* To assess the safety and tolerability of a daily single oral dose of 20 mg tasimelteon.

DETAILED DESCRIPTION:
REM behavior disorder (RBD) is characterized by abnormal behaviors that emerge from REM sleep and can lead to injury and disturbed sleep. Most patients have frequent events - typically more than once per week. Abnormalities can be seen almost nightly and consist of intermittent loss of the normal atonia of REM sleep. This phenomenon is used as diagnostic criterion even in the absence of an overt clinical event during the night.

RBD has serious consequences for the health of the patient. Besides risk of sometimes severe injury, a direct consequence of a violent nocturnal movement, it often leads to sleep disruption. Furthermore, it is commonly seen in association with Parkinson's disease and many experts in the field consider it a prodrome of neurodegenerative conditions. Other comorbidities may include a higher risk of cerebral hemorrhage as well as stroke. Multiple factors may contribute to the risk of RBD. Aside from neurodegenerative conditions, RBD is seen in association with disorders of REM sleep regulations: narcolepsy, post-traumatic stress disorder, or with use of selective serotonin reuptake inhibitors (SSRIs).

In healthy individuals, REM sleep is closely linked to circadian phase, with a peak a little after the nadir of the core body temperature, and thus also around the time when melatonin secretion is maximal. Studies using a forced desynchrony protocol suggest that the circadian system has a primary effect of REM sleep regulation with a modifying effect from the homeostatic factors. Various other factors affect REM sleep, including complex interactions with the serotonergic system, primarily from the raphe nuclei in the medulla, which inhibit the REM generating pontine tegmentum nuclei. Clinically, patients treated with antidepressants, particularly with serotononergic properties (particularly SSRIs), tend to suppress REM sleep and may also lead to REM without atonia and/or trigger RBD events.

The melatonin MT1 and MT2 receptors likely both affect the NREM/REM ratio with activation of the MT2 leading to earlier and more abundant NREM sleep, while MT1 receptors favoring REM sleep. Furthermore, RBD is common in patients with Parkinson's disease, and a reduced number of melatonin receptors have been found in the areas involved in the neurodegeneration: a recent study found a reduced number of MT1 receptor expression in the striatum and amygdala, and a reduced MT2 receptor expression in the substantia nigra and amygdala. In addition to circadian phase shift, activation of melatonin MT1 and MT2 receptors has been implicated as a potential protective mechanism against multiple other progressive neurodegenerative disorders, while MT2 receptors have been implicated in neurogenesis. Thus, REM suppression and/or disruption, as a result of the neurodegenerative process, that also involves impaired MT1 and MT2 receptor function may be a key mechanism for RBD pathophysiology and potential therapeutic target.

Treatment options for RBD are limited. The most commonly used agent is clonazepam, which has to be used in caution in patient with dementia symptoms and has many potentially serious side effects. Due to the strong association with neurodegenerative conditions, RBD patients are likely to have contraindications for benzodiazepine treatment. This creates a need for other medications that can be safely used in patients who are elderly and/or have neurodegenerative comorbid conditions. If the mechanism for RBD include REM sleep disruption, can improved REM sleep regulation lead to a better treatment? Melatonin is the most common therapeutic alternative to clonazepam for RBD. Initial studies may have been partially prompted by its high clinical convenience: a very favorable side effect profile, and availability in the US. It was first reported as effective in a case report in 1997, of a 64 year old man who experienced improvement of his RBD symptoms after treatment with 3 mg melatonin, without any change in his REM proportion on polysomnography. Further studies have included open label case series. In one recent study, melatonin was found to be equally effective as clonazepam for RBD treatment. However, studies have been small, open label, sometimes retrospective, and generally the timing of melatonin is not consistently reported.

Use of melatonin has a number of clinical challenges, since the medication is over the counter, not regulated, and dose and bioavailability can vary widely. Can melatonin agonists, which have a higher affinity to melatonin receptors also be used for treatment? Indeed, ramelteon has been reported successful in some cases. In 2013, Nomura et al used ramelteon, 8 mg in two patients who had polysomnographically confirmed RBD in association with parkinsonian syndromes. One of them had multisystem atrophy, and could not tolerate clonazepam due to the lability of her blood pressure, and the other had persistent symptoms despite clonazepam treatment. Both individuals had improvement of their RBD symptoms, including the RBD severity scale (RBDSS). Later Esaki et al treated 12 consecutive patients with idiopathic RBD in an open label trial, using 8 mg ramelteon given 30 minutes before bedtime and reported a trend towards improvement. Yet another study examined the effect of ramelteon on motor and non-motor symptoms in patients with Parkinson's disease, with or without RBD, and reported improvement in a variety of measures after treatment, including a statistically significant RBD improvement.

Novel data has emerged in the past two years regarding the chronotherapeutic aspects of RBD, suggesting that a potential not only for improved symptom control, but also long-term benefit in terms of decreasing neurodegeneration.

However, due to a large first pass effect, the mean systemic availability of ramelteon following an oral dose is less than 2%, and there is a large degree of inter-subject variability in plasma concentration after exposure. Thus, another melatonin agonist could be very helpful for patients with REM behavior disorder, potentially providing a more effective treatment option for this disease, and allowing safer control of the symptoms for those who cannot use benzodiazepines. A potent activator of the MT1 receptors, such as tasimelteon, could be an ideal RBD treatment. To better evaluate this important clinical question, I propose to evaluate the efficacy of tasimelteon as a potential treatment for RBD.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of REM sleep behavior disorder, confirmed polysomnography
2. Ability to participate in the trial

Exclusion criteria:

1. Contraindication to tasimelteon
2. medical or psychiatric conditions that limit ability to participate or increase risk to the individual

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Daily Sleep Diary - Visual Fill-In | Daily for 8 weeks (both baseline and treatment phases)
  The daily sleep diary contains a diagram similar to a calendar that the participant can track their intake of caffeine, medicine, and alcohol, if they exercised, when they went to bed, fell asleep, or took a nap, and when they woke up. All recordings will be measured as number of events/time of day.
Daily Sleep Diary - Time Keeping | Daily for 8 weeks (both baseline and treatment phases)
  The daily sleep diary also contains a series of questions. Some of them ask the participant to record the time the diary is completed, the time they took the study drug, and the time that they think they had a dream reenactment event. All of these will be recorded in 24:00 format.
Daily Sleep Diary - Sleep Questions | Daily for 8 weeks (both baseline and treatment phases)
  The daily sleep diary also asks participants subjective questions like did you sleep last night, did you wake up naturally, and did you take the study drug last night? These will be recorded as yes/no responses.
Daily Sleep Diary - Dream Enactment | Daily for 8 weeks (both baseline and treatment phases)
  The daily sleep diary also asks participants to recall how many dream enactments they had the previous night if any at all. This will be recorded as a numerical value.

SECONDARY OUTCOMES:
Clinical Global Impression of Change | 1 Month after study
  Investigator-rated Assessment of Global Improvement in participant symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Milena Pavlova, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haba-Rubio J, Frauscher B, Marques-Vidal P, Toriel J, Tobback N, Andries D, Preisig M, Vollenweider P, Postuma R, Heinzer R. Prevalence and determinants of rapid eye movement sleep behavior disorder in the general population. Sleep. 2018 Feb 1;41(2):zsx197. doi: 10.1093/sleep/zsx197. PMID 29216391
- [Background] Chiu HF, Wing YK, Lam LC, Li SW, Lum CM, Leung T, Ho CK. Sleep-related injury in the elderly--an epidemiological study in Hong Kong. Sleep. 2000 Jun 15;23(4):513-7. PMID 10875558
- [Background] Boeve BF, Molano JR, Ferman TJ, Lin SC, Bieniek K, Tippmann-Peikert M, Boot B, St Louis EK, Knopman DS, Petersen RC, Silber MH. Validation of the Mayo Sleep Questionnaire to screen for REM sleep behavior disorder in a community-based sample. J Clin Sleep Med. 2013 May 15;9(5):475-80. doi: 10.5664/jcsm.2670. PMID 23674939
- [Background] Stiasny-Kolster K, Mayer G, Schafer S, Moller JC, Heinzel-Gutenbrunner M, Oertel WH. The REM sleep behavior disorder screening questionnaire--a new diagnostic instrument. Mov Disord. 2007 Dec;22(16):2386-93. doi: 10.1002/mds.21740. PMID 17894337
- [Background] Postuma RB, Gagnon JF, Montplaisir J. Rapid eye movement sleep behavior disorder as a biomarker for neurodegeneration: the past 10 years. Sleep Med. 2013 Aug;14(8):763-7. doi: 10.1016/j.sleep.2012.09.001. Epub 2012 Oct 8. PMID 23058689
- [Background] Marion MH, Qurashi M, Marshall G, Foster O. Is REM sleep behaviour disorder (RBD) a risk factor of dementia in idiopathic Parkinson's disease? J Neurol. 2008 Feb;255(2):192-6. doi: 10.1007/s00415-008-0629-9. Epub 2008 Jan 29. PMID 18217187
- [Background] Ma C, Pavlova M, Liu Y, Liu Y, Huangfu C, Wu S, Gao X. Probable REM sleep behavior disorder and risk of stroke: A prospective study. Neurology. 2017 May 9;88(19):1849-1855. doi: 10.1212/WNL.0000000000003902. Epub 2017 Apr 7. PMID 28389588
- [Background] Nightingale S, Orgill JC, Ebrahim IO, de Lacy SF, Agrawal S, Williams AJ. The association between narcolepsy and REM behavior disorder (RBD). Sleep Med. 2005 May;6(3):253-8. doi: 10.1016/j.sleep.2004.11.007. PMID 15854856
- [Background] Boeve BF. REM sleep behavior disorder: Updated review of the core features, the REM sleep behavior disorder-neurodegenerative disease association, evolving concepts, controversies, and future directions. Ann N Y Acad Sci. 2010 Jan;1184:15-54. doi: 10.1111/j.1749-6632.2009.05115.x. PMID 20146689
- [Background] Czeisler CA, Zimmerman JC, Ronda JM, Moore-Ede MC, Weitzman ED. Timing of REM sleep is coupled to the circadian rhythm of body temperature in man. Sleep. 1980;2(3):329-46. PMID 7403736
- [Background] Dijk DJ, Czeisler CA. Contribution of the circadian pacemaker and the sleep homeostat to sleep propensity, sleep structure, electroencephalographic slow waves, and sleep spindle activity in humans. J Neurosci. 1995 May;15(5 Pt 1):3526-38. doi: 10.1523/JNEUROSCI.15-05-03526.1995. PMID 7751928
- [Background] Carskadon MA, Dement WC. Sleep studies on a 90-minute day. Electroencephalogr Clin Neurophysiol. 1975 Aug;39(2):145-55. doi: 10.1016/0013-4694(75)90004-8. PMID 50211
- [Background] Lee K, Baron K, Soca R, Attarian H. The Prevalence and Characteristics of REM Sleep without Atonia (RSWA) in Patients Taking Antidepressants. J Clin Sleep Med. 2016 Mar;12(3):351-5. doi: 10.5664/jcsm.5582. PMID 26446247
- [Background] Arnaldi D, Fama F, De Carli F, Morbelli S, Ferrara M, Picco A, Accardo J, Primavera A, Sambuceti G, Nobili F. The Role of the Serotonergic System in REM Sleep Behavior Disorder. Sleep. 2015 Sep 1;38(9):1505-9. doi: 10.5665/sleep.5000. PMID 25845692
- [Background] Liu J, Clough SJ, Hutchinson AJ, Adamah-Biassi EB, Popovska-Gorevski M, Dubocovich ML. MT1 and MT2 Melatonin Receptors: A Therapeutic Perspective. Annu Rev Pharmacol Toxicol. 2016;56:361-83. doi: 10.1146/annurev-pharmtox-010814-124742. Epub 2015 Oct 23. PMID 26514204
- [Background] Adi N, Mash DC, Ali Y, Singer C, Shehadeh L, Papapetropoulos S. Melatonin MT1 and MT2 receptor expression in Parkinson's disease. Med Sci Monit. 2010 Feb;16(2):BR61-7. PMID 20110911
- [Background] Dubocovich ML, Markowska M. Functional MT1 and MT2 melatonin receptors in mammals. Endocrine. 2005 Jul;27(2):101-10. doi: 10.1385/ENDO:27:2:101. PMID 16217123
- [Background] Lee CH, Yoo KY, Choi JH, Park OK, Hwang IK, Kwon YG, Kim YM, Won MH. Melatonin's protective action against ischemic neuronal damage is associated with up-regulation of the MT2 melatonin receptor. J Neurosci Res. 2010 Sep;88(12):2630-40. doi: 10.1002/jnr.22430. PMID 20544829
- [Background] Kunz D, Bes F. Melatonin effects in a patient with severe REM sleep behavior disorder: case report and theoretical considerations. Neuropsychobiology. 1997;36(4):211-4. doi: 10.1159/000119383. PMID 9396020
- [Background] Takeuchi N, Uchimura N, Hashizume Y, Mukai M, Etoh Y, Yamamoto K, Kotorii T, Ohshima H, Ohshima M, Maeda H. Melatonin therapy for REM sleep behavior disorder. Psychiatry Clin Neurosci. 2001 Jun;55(3):267-9. doi: 10.1046/j.1440-1819.2001.00854.x. PMID 11422870
- [Background] Boeve BF, Silber MH, Ferman TJ. Melatonin for treatment of REM sleep behavior disorder in neurologic disorders: results in 14 patients. Sleep Med. 2003 Jul;4(4):281-4. doi: 10.1016/s1389-9457(03)00072-8. PMID 14592300
- [Background] Kunz D, Bes F. Melatonin as a therapy in REM sleep behavior disorder patients: an open-labeled pilot study on the possible influence of melatonin on REM-sleep regulation. Mov Disord. 1999 May;14(3):507-11. doi: 10.1002/1531-8257(199905)14:33.0.co;2-8. PMID 10348479
- [Background] McGrane IR, Leung JG, St Louis EK, Boeve BF. Melatonin therapy for REM sleep behavior disorder: a critical review of evidence. Sleep Med. 2015 Jan;16(1):19-26. doi: 10.1016/j.sleep.2014.09.011. Epub 2014 Oct 13. PMID 25454845
- [Background] Nomura T, Kawase S, Watanabe Y, Nakashima K. Use of ramelteon for the treatment of secondary REM sleep behavior disorder. Intern Med. 2013;52(18):2123-6. doi: 10.2169/internalmedicine.52.9179. PMID 24042525
- [Background] Esaki Y, Kitajima T, Koike S, Fujishiro H, Iwata Y, Tsuchiya A, Hirose M, Iwata N. An Open-Labeled Trial of Ramelteon in Idiopathic Rapid Eye Movement Sleep Behavior Disorder. J Clin Sleep Med. 2016 May 15;12(5):689-93. doi: 10.5664/jcsm.5796. PMID 26857053
- [Background] Kashihara K, Nomura T, Maeda T, Tsuboi Y, Mishima T, Takigawa H, Nakashima K. Beneficial Effects of Ramelteon on Rapid Eye Movement Sleep Behavior Disorder Associated with Parkinson's Disease - Results of a Multicenter Open Trial. Intern Med. 2016;55(3):231-6. doi: 10.2169/internalmedicine.55.5464. Epub 2016 Feb 1. PMID 26831015
- [Background] Rajaratnam SM, Polymeropoulos MH, Fisher DM, Roth T, Scott C, Birznieks G, Klerman EB. Melatonin agonist tasimelteon (VEC-162) for transient insomnia after sleep-time shift: two randomised controlled multicentre trials. Lancet. 2009 Feb 7;373(9662):482-91. doi: 10.1016/S0140-6736(08)61812-7. Epub 2008 Dec 4. PMID 19054552
- [Background] Postuma RB, Arnulf I, Hogl B, Iranzo A, Miyamoto T, Dauvilliers Y, Oertel W, Ju YE, Puligheddu M, Jennum P, Pelletier A, Wolfson C, Leu-Semenescu S, Frauscher B, Miyamoto M, Cochen De Cock V, Unger MM, Stiasny-Kolster K, Fantini ML, Montplaisir JY. A single-question screen for rapid eye movement sleep behavior disorder: a multicenter validation study. Mov Disord. 2012 Jun;27(7):913-6. doi: 10.1002/mds.25037. Epub 2012 May 30. PMID 22729987